CLINICAL TRIAL: NCT01998048
Title: Operative Treatment of Traumatic Anteroinferior Shoulder Instability in Young Male Patients. The Outcome of Arthroscopic Bankart vs. Open Latarjet Stabilization Surgery, a Randomized Controlled Trial.
Brief Title: Operative Treatment of Traumatic Anteroinferior Shoulder Instability in Young Male Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Ville Aarimaa, adjunct professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FINNISH
Record Dates: First submitted 2013-11-24; First posted 2013-11-28 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Shoulder Instability
Keywords: surgical treatment; Bankart; Latarjet; redislocation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Latarjet (Active Comparator): 60 patients treated with open Latarjet operation
  Interventions: Procedure: Latarjet
- Bankart (Active Comparator): 60 patients treated with arthroscopic Bankart operation
  Interventions: Procedure: Bankart

INTERVENTIONS:
Procedure: Latarjet — A diagnostic arthroscopy is performed before the Latarjet operation in general anaesthesia. In case of a significant Hill-Sachs defect an additional remplissage procedure may be performed according to surgeons' decision by inserting 1 to 2 more suture anchors according to surgeon's preference into the deepest portion of the Hill-Sachs defect and tying the infraspinatus tendon down to fill the bony defect. Thereafter an open Latarjet operation is performed using standard techniques described by Walch or de Beer. A deltopectoral incision is used. The coracoid process is osteotomized and ventrally prepared to bleeding bone. The coracoid process is then transferred through the middle of the subscapularis and re-attached on to the freshened neck of the glenoid, just medial to the joint line with two screws and washers, according to the surgeon's preference.
  Arms: Latarjet
Procedure: Bankart — An arthroscopic Bankart operation is performed in general anaesthesia according to current practise (Provencher 2010). The intra-articular findings are recorded and the anteroinferior labrum and the IGHL are mobilized until subscapular muscle fibers can be seen. The IGHL complex is then re-attached to the freshened neck of the glenoid with 2 to 3 suture anchors according to surgeon's preference to re-create labral bumper and capsular tension. In case of a significant Hill-Sachs defect an additional remplissage procedure may be performed according to surgeon's decision by inserting 1 to 2 more suture anchors, according to surgeon's preference into the deepest portion of the Hill-Sachs defect and tying the infraspinatus tendon down to fill the bony defect.
  Arms: Bankart

SUMMARY:
Glenohumeral joint is prone to instability, i.e. the humeral head may dislocate off the scapular glenoid plate especially in the anteroinferior direction. Surgical treatment of shoulder instability aims at restoration of shoulder stability. The purpose of this trial is to investigate the difference in outcome after arthroscopic Bankart operation compared with open Latarjet operation in the treatment of a residual instability after a traumatic primary dislocation in young males.

ELIGIBILITY:
Inclusion Criteria:

1. Subluxation or fear of shoulder dislocation after a previous, reduced and primarily conservatively treated (for more than 3 months) traumatic anteroinferior shoulder dislocation, or redislocation after a primary shoulder dislocation.
2. Clinically documented anteroinferior instability (ie. a positive apprehension and relocation test (Jobe)).
3. X-ray (true ap, 30 degrees oblique ap, Y- and axillary projections), 2- and 3-dimensional computed tomography (2D and 3D CT) and magnetic resonance imaging arthrography (MRA) documentation of the joint.
4. Congruency of the shoulder joint on imaging investigations.
5. Young adult male patient 16-25 years of age (15 years < patient < 26 years ).
6. Patient's willingness for operative treatment.
7. Written informed consent from participating subject.

Exclusion Criteria:

1. Non-congruency of the glenohumeral joint on imaging investigations.
2. Concomitant dislocated fractures (requiring operative treatment) of the humerus or the scapula (other than Hill-Sachs lesion or bony Bankart lesion)
3. Severe grade 2 or above (Samilson et Prieto) osteoarthrosis of the glenohumeral joint detected in X-ray investigation.
4. A humeral avulsion of glenohumeral ligaments (HAGL) detected in MRA investigation.
5. Concomitant ipsilateral plexus or axillar nerve injury affecting motor function.
6. Life threatening other concomitant injuries (i.e. multitrauma patient).
7. Stiffness of the glenohumeral joint (restricted passive external rotation less than 30 degrees measured in standing position, arm at side).
8. Age under 16 or above 25 years.
9. Open physis with significant growth expectation.
10. Intellectual disability, history of seizures with high risk of recurrence, existing significant malignant, haematological, endocrine, metabolic, or rheumatoid disease.

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
recurrence of instability | 5 years
  The recurrence of instability (re-dislocation, subluxation, positive apprehension) is used as a primary outcome measure together with WOSI score two and five years postoperatively.

OTHER OUTCOMES:
shoulder state | 5 years
  Secondary outcome measures include: level and intensity to perform sports activities, subjective visual analogue estimation of the shoulder condition, Constant score, Oxford score, and SSV.

CONTACTS AND LOCATIONS:
Overall Officials: Ville Äärimaa, Adjunct Professor, Principal Investigator — Turku University Hospital
Locations (8):
- Finland (8):
  - Helsinki University Hospital, Helsinki
  - Keski-Suomen keskussairaala, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Satakunnan keskussairaala, Pori
  - Hatanpään sairaala, Tampere
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Kukkonen J, Elamo S, Flinkkila T, Paloneva J, Mantysaari M, Joukainen A, Lehtinen J, Lepola V, Holstila M, Kauko T, Aarimaa V; FINNISH (Finnish Instability Shoulder Study) Investigators. Arthroscopic Bankart versus open Latarjet as a primary operative treatment for traumatic anteroinferior instability in young males: a randomised controlled trial with 2-year follow-up. Br J Sports Med. 2022 Mar;56(6):327-332. doi: 10.1136/bjsports-2021-104028. Epub 2021 Sep 22. PMID 34551902